CLINICAL TRIAL: NCT01239732
Title: Global Study to Assess the Addition of Bevacizumab to Carboplatin and Paclitaxel as Front-line Treatment of Epithelial Ovarian Cancer, Fallopian Tube Carcinoma or Primary Peritoneal Carcinoma
Brief Title: A Study of the Addition of Avastin (Bevacizumab) to Carboplatin and Paclitaxel Therapy in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO22923; 2010-019525-34 (EudraCT Number)
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Bevacizumab; Carboplatin

ARMS (1):
- Bevacizumab + Paclitaxel + Carboplatin (Experimental): Participants will receive bevacizumab 15 mg/kg IV on Day 1 every 3 weeks from Cycle 1 to Cycle 36 (initially concurrent with chemotherapy, then continued as a single agent following the completion of chemotherapy), or until protocol defined disease progression or until unacceptable toxicity (whichever occurred first). Participants will receive paclitaxel 175 mg/m^2 IV on Day 1 every 3 weeks or 80 mg/m^2 IV every week and carboplatin (AUC 5-6) IV on Day 1 every 3 weeks for a minimum of 4 and maximum of 8 cycles (including up to 4 pre-surgical cycles), or until protocol defined disease progression, or unacceptable toxicity (whichever occurred first).
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel — 175 mg/m^2 on Day 1 every 3 weeks or at a dose of 80 mg/m^2 every week for a minimum of 4 cycles and not more than 8 cycles or until disease progression or unacceptable toxicity, whichever occurs first
Drug: Bevacizumab — 15 mg/kg intravenously on Day 1 of every cycle for up to 36 cycles of 3 weeks each or until disease progression or unacceptable toxicity, whichever occurs first
  Other Names: Avastin
Drug: Carboplatin — AUC 5-6 mg/ml/min on Day 1 every 3 weeks for a minimum of 4 cycles and not more than 8 cycles or until disease progression or unacceptable toxicity, whichever occurs first

SUMMARY:
This open-label, non-comparative, multi-center study will assess the safety profile and efficacy of Avastin (bevacizumab) when added to carboplatin and paclitaxel therapy in participants with epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma. Participants will receive 15 milligrams/kilogram (mg/kg) Avastin intravenously (IV) on Day 1 of every cycle for up to 36 cycles of 3 weeks each, carboplatin (area under the plasma concentration-time curve [AUC] 5-6 mg/ml/min) on Day 1 every 3 weeks for a maximum of 8 cycles and paclitaxel 175 milligram per square meter (mg/m^2) on Day 1 every 3 weeks or 80 mg/m^2 every week for a maximum of 8 cycles. The anticipated time on study drug will be 108 weeks or until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian carcinoma, fallopian tube carcinoma, primary peritoneal carcinoma or clear cell carcinoma or carcinosarcoma. Participants with recurrent ovarian cancer who have been previously treated with surgery alone for their early stage disease are eligible.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0, 1 or 2
* Life expectancy greater than or equal to (>=3) months

Exclusion Criteria:

* Participants with non-epithelial ovarian cancer, ovarian tumors with low malignant potential (i.e., borderline tumors), or synchronous primary endometrial carcinoma
* Previous systemic therapy for ovarian cancer. Prior neo-adjuvant chemotherapy is allowed
* Planned intraperitoneal cytotoxic chemotherapy
* Radiotherapy within 28 days of Day 1, Cycle 1
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to first dose of Avastin
* History or evidence of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade >=1 arterial thromboembolic event or Grade >=3 venous thromboembolic event within 6 months prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2010-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (199):
- Argentina (3):
  - Buenos Aires
  - Rosario
  - San Miguel de Tucumán
- Austria (7):
  - Graz
  - Innsbruck
  - Ried-innkreis
  - Salzburg
  - Steyr
  - Vienna
  - Villach
- Brazil (8):
  - Fortaleza, Ceará
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Piracicaba, São Paulo
  - São Paulo, São Paulo
- Bulgaria (3):
  - Sofia
  - Varna
  - Veliko Tarnovo
- Canada (5):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Denmark (3):
  - Aalborg
  - Roskilde
  - Vejle
- Egypt (2):
  - Cairo
  - Tanta
- Estonia (2):
  - Tallinn
  - Tartu
- France (15):
  - Amiens
  - Bordeaux
  - Brest
  - Caen
  - Clermont-Ferrand
  - Grenoble
  - Lille
  - Lyon
  - Marseille
  - Mougins
  - Paris
  - Reims
  - Strasbourg
  - Toulouse
  - Villejuif
- Greece (5):
  - Athens
  - Heraklion, Crete
  - Larissa
  - Pátrai
  - Thessaloniki
- Hong Kong, Hong Kong
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
- India (6):
  - Bangalore
  - Hyderabad
  - Jaipur
  - Kochi
  - New Delhi
  - Pune
- Dublin, Ireland
- Israel (10):
  - Afula
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Italy (16):
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Meldola, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Brescia, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Saronno, Lombardy
  - Novara, Piedmont
  - Turin, Piedmont
  - Palermo, Sicily
  - Florence, Tuscany
  - Pisa, Tuscany
  - Perugia, Umbria
  - Terni, Umbria
- Ash Shuwaykh, Kuwait
- Latvia (2):
  - Daugavpils
  - Riga
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Mexico (3):
  - Distrito Federal
  - Oaxaca City
  - Toluca
- Netherlands (14):
  - Alkmaar
  - Amsterdam
  - Apeldoorn
  - Blaricum
  - Breda
  - Capelle aan den IJssel
  - Deventer
  - Dordrecht
  - Eindhoven
  - Leidschendam
  - Rotterdam
  - Sittard-Geleen
  - The Hague
  - Utrecht
- North Macedonia (2):
  - Bitola
  - Skopje
- Poland (2):
  - Bydgoszcz
  - Warsaw
- Porto, Portugal
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Iași
- Russia (6):
  - Barnaul
  - Moscow
  - Obninsk, Kaluzhskaya Region
  - Saint Petersburg
  - Stavropol
  - Ufa
- Dammam, Saudi Arabia
- Serbia (2):
  - Belgrade
  - Niš
- Slovakia (2):
  - Bratislava
  - Košice
- Slovenia (2):
  - Ljubljana
  - Maribor
- South Africa (3):
  - Durban
  - Johannesburg
  - Sandton
- Spain (43):
  - Albacete, Albacete
  - Alicante, Alicante
  - Elda, Alicante
  - Badajoz, Badajoz
  - Llerena (Badajoz), Badajoz
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Manresa, Barcelona
  - Burgos, Burgos
  - Cáceres, Caceres
  - Cadiz, Cadiz
  - Jerez de la Frontera, Cadiz
  - Castellon, Castellon
  - Ciudad Real, Ciudad Real
  - Córdoba, Cordoba
  - Girona, Girona
  - Granada, Granada
  - Guadalajara, Guadalajara
  - Donostia / San Sebastian, Guipuzcoa
  - San Sebastián de los Reyes, Guipuzcoa
  - Jaén, Jaen
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Las Palmas de Gran Canaria, Las Palmas
  - Lugo, Lugo
  - Leganés, Madrid
  - Madrid, Madrid
  - Málaga, Malaga
  - Navarra, Navarre
  - Oviedo, Principality of Asturias
  - Salamanca, Salamanca
  - Segovia, Segovia
  - Seville, Sevilla
  - Reus, Tarragona
  - San Cristóbal de La Laguna, Tenerife
  - Santa Cruz de Tenerife, Tenerife
  - Toledo, Toledo
  - San Juan, Valencia
  - Valencia, Valencia
  - Valladolid, Valladolid
  - Barakaldo, Vizcaya
  - Bilbao, Vizcaya
  - Zaragoza, Zaragoza
- Sweden (6):
  - Eskilstuna
  - Falun
  - Karlstad
  - Örebro
  - Umeå
  - Uppsala
- Switzerland (6):
  - Aarau
  - Baden
  - Bellinzona
  - Bern
  - Geneva
  - Zurich
- Taiwan (2):
  - Taipei
  - Taoyuan Hsien
- Turkey (Türkiye) (3):
  - Ankara
  - Diyarbakır
  - Istanbul
- Montevideo, Uruguay

REFERENCES:
- [Derived] Oza AM, Selle F, Davidenko I, Korach J, Mendiola C, Pautier P, Chmielowska E, Bamias A, DeCensi A, Zvirbule Z, Gonzalez-Martin A, Hegg R, Joly F, Zamagni C, Gadducci A, Martin N, Robb S, Colombo N. Efficacy and Safety of Bevacizumab-Containing Therapy in Newly Diagnosed Ovarian Cancer: ROSiA Single-Arm Phase 3B Study. Int J Gynecol Cancer. 2017 Jan;27(1):50-58. doi: 10.1097/IGC.0000000000000836. PMID 27749456

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study has been completed. However, the efficacy and safety results up to the clinical database cutoff date of 07 December 2014 are provided.
Groups:
- Bevacizumab + Paclitaxel + Carboplatin: Participants received bevacizumab 15 milligrams/kilogram (mg/kg) intravenously (IV) on Day 1 every 3 weeks from Cycle 1 (1 cycle = 3 weeks) to Cycle 36 (initially concurrent with chemotherapy, then continued as a single agent following the completion of chemotherapy), or until protocol-defined disease progression or until unacceptable toxicity (whichever occurred first). The 15 mg/kg dose every 3 weeks was the recommended dose; however a dose of IV bevacizumab 7.5 mg/kg every 3 weeks was permissible, but was to be selected prior to the first dosing of bevacizumab. Participants received paclitaxel 175 milligram per square meter (mg/m^2) IV on Day 1 every 3 weeks or 80 mg/m^2 IV every week and carboplatin (area under the plasma concentration-time curve [AUC] 5-6) IV on Day 1 every 3 weeks for a minimum of 4 and maximum of 8 cycles (including up to 4 pre-surgical cycles), or until protocol-defined disease progression, or unacceptable toxicity (whichever occurred first).
Period: Overall Study
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Started | 1021
Completed | 0
Not Completed | 1021
Not completed — Termination of study per protocol | 667
Not completed — Death | 226
Not completed — Withdrawal by Subject | 87
Not completed — Adverse Event | 6
Not completed — Protocol Violation | 3
Not completed — Participant non compliance | 5
Not completed — Study termination by sponsor | 2
Not completed — Investigator's decision | 4
Not completed — Treatment failure | 2
Not completed — Other | 19

BASELINE CHARACTERISTICS:
Population: Safety population: included all participants who received at least one dose of study medication.
Groups:
- Bevacizumab + Paclitaxel + Carboplatin: Participants received bevacizumab 15 mg/kg IV on Day 1 every 3 weeks from Cycle 1 (1 cycle = 3 weeks) to Cycle 36 (initially concurrent with chemotherapy, then continued as a single agent following the completion of chemotherapy), or until protocol-defined disease progression or until unacceptable toxicity (whichever occurred first). The 15 mg/kg dose every 3 weeks was the recommended dose; however a dose of IV bevacizumab 7.5 mg/kg every 3 weeks was permissible, but was to be selected prior to the first dosing of bevacizumab. Participants received paclitaxel 175 mg/m^2 IV on Day 1 every 3 weeks or 80 mg/m^2 IV every week and carboplatin (AUC 5-6) IV on Day 1 every 3 weeks for a minimum of 4 and maximum of 8 cycles (including up to 4 pre-surgical cycles), or until protocol-defined disease progression, or unacceptable toxicity (whichever occurred first).
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 1021
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1021
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Day 1 up to 30 days after last dose of study treatment (until data cutoff 07 December 2014, up to 4 years)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 1021
percentage of participants | 97.8

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time between the date of first administration of any study treatment and the date of first documented protocol-defined disease progression (that is [i.e.], radiologically by Response Evaluation Criteria In Solid Tumors [RECIST], clinical, or symptomatic) or death, whichever occurred first. Participants who had neither progressed nor died at the time of data cut-off (07 December 2014), or participants who were withdrawn from study, or lost to follow-up without documented progression, were censored. Kaplan-Meier estimation was used for median time to PFS.
Time Frame: Day 1, at end of Cycles 3 and 6, then every 6 cycles while receiving bevacizumab, and then at bevacizumab cessation, every 26 weeks after cessation of bevacizumab until disease progression or death until data cutoff 07 December 2014, up to 4 years
Population: Intent to treat population included all participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 1021
months | 25.5 [23.7 to 27.6]

3. Secondary Outcome: Percentage of Participants Achieving Best Overall Response of Complete Response (CR) or Partial Response (PR) According to RECIST Version 1.0
Description: Best overall response (BOR) according to RECIST Version 1.0 was categorized as: CR, PR, progressive disease (PD), stable disease (SD). CR: disappearance of all target lesions and non-target lesions. PR: >=30% decrease in sum of the longest diameters (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non-target lesions. PD: Natural progression or deterioration of the malignancy under study (including new sites of metastasis). SD: neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started. Participants with a BOR of CR and PR were defined as responders, while participants with a BOR of SD, PD, or unable to assess were defined as non-responders.
Time Frame: Day 1, at end of Cycles 3 and 6, then every 6 cycles while receiving bevacizumab, and then at bevacizumab cessation, every 26 weeks (Q26W) after cessation of bevacizumab until disease progression or death until data cutoff 07 December 2014, up to 4 years
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 421
percentage of participants | 72.7 [68.2 to 76.9]

4. Secondary Outcome: Percentage of Participants Achieving an Overall Response by 50% Carcinoma Antigen 125 (CA-125) Response Criteria
Description: CA-125 responders: Participants with the value of CA-125 reduced by at least 50% and confirmed with a consecutive CA-125 assessment performed at an interval of at least 28 days. Overall response according to CA-125 was only evaluated for participants with a pre-treatment CA-125 within 3 days prior to start of any study treatment of at least twice the upper limit of normal (ULN).
Time Frame: 3 days prior to Day 1 of every cycle, then every 6 weeks (Q6W) during the first year, every 3 months (Q3M) in the second and third year, every 6 months (Q6M) in the fourth year of the study (until data cutoff 07 December 2014, up to 4 years)
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 340
percentage of participants | 91.8 [88.3 to 94.5]

5. Secondary Outcome: Percentage of Participants Achieving an Overall Response by RECIST Version 1.0 and/or 50% CA-125 Response Criteria
Description: Overall response was only evaluated for participants who were evaluable according to RECIST v1.0 with a measurable disease at baseline and/or according to CA-125 with a pre-treatment CA-125 within 3 days prior to start of any study treatment of at least twice the ULN. RECIST responders: Participants achieving an overall response of CR (disappearance of all target lesions and non-target lesions) or PR (>=30% decrease in sum of the LD of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non target lesions). CA-125 responders: Participants with the value of CA-125 reduced by at least 50% and confirmed with a consecutive CA-125 assessment performed at an interval of at least 28 days.
Time Frame: RECIST: Day 1, at end of Cycles 3 and 6, then every 6 cycles, at bevacizumab cessation, Q26W after cessation; CA-125: 3 days before Day 1 of every cycle, then Q6W(1st year), Q3M(2nd-3rd year), Q6M(4th year); until data cutoff 07Dec2014, up to 4 years
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 578
percentage of participants | 82.4 [79.0 to 85.4]

6. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR was defined as the time from the first documented response (CR or PR per RECIST v1.0), to the first documented protocol-defined disease progression (i.e., radiologically by RECIST, clinical, or symptomatic) or death, whichever occurred first. Participants who had neither progressed nor died at the time of data cut-off (07 December 2014), or participants who were withdrawn from study, or lost to follow-up without documented progression, were censored. RECIST responders: Participants achieving an overall response of CR (disappearance of all target lesions and non-target lesions) or PR (>=30% decrease in sum of the LD of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non-target lesions). Disease progression: Natural progression or deterioration of the malignancy under study (including new sites of metastasis).
Time Frame: as for outcome 2
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 1021
months | 18.2 [16.6 to 19.6]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first administration of any study treatment to the date of death, regardless of the cause of death. Participants without the event of death were censored at the last date in the study, defined as the latest date of the following: the date of first administration of study treatment, date of last study treatment, date of last visit, or date last known to be alive. Kaplan-Meier estimation was used for OS.
Time Frame: First administration of any study treatment until death or data cutoff 07 December 2014, up to 4 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 1021
months | NA [NA to NA] — The median and 95% confidence interval were not calculable because less than 50% of participants had the event.

8. Secondary Outcome: Biological Progression-free Interval
Description: Biological progression-free interval is defined as the interval from the date of the first administration of any study treatment to the date of the first documented serial elevation of the ovarian cancer mucin CA-125. More precisely, this is defined as the first documented increase in CA-125 levels as follows: (1) CA-125 greater than or equal to 2 times the upper level of normal (ULN) on 2 occasions at least 1 week apart (for participants with CA-125 within normal range pre-treatment) or (2) CA-125 greater than or equal to 2 times the ULN on 2 occasions at least 1 week apart (for participants with elevated CA-125 pre-treatment and initial normalization of CA-125 on-treatment) or (3) CA-125 greater than or equal to 2 times the nadir value, which is the lowest observed CA-125 value per participant on 2 occasions at least 1 week apart (for participants with elevated CA-125 pre-treatment which never normalized).
Time Frame: 3 days prior to Day 1 of every cycle, then every 6 weeks during the first year, every 3 months in the second and third year, every 6 months in the fourth year of the study (until data cutoff 07 December 2014, up to 4 years)
Population: Previous studies linking CA-125 levels with bevacizumab exposure as a potential secondary outcome measure for PFS did not produce any reliable information. Therefore, it was decided that data for this outcome measure should not be analyzed, as agreed with the study steering committee.
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after last dose of study treatment (until data cutoff 07 December 2014, up to 4 years)
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 285/1021
Other Adverse Events (participants affected / at risk) | 980/1021
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel + Carboplatin (N=1021)
Diarrhoea (Gastrointestinal disorders) | 13
Intestinal obstruction (Gastrointestinal disorders) | 11
Ileus (Gastrointestinal disorders) | 9
Subileus (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 8
Small intestinal obstruction (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Gastrointestinal perforation (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Umbilical hernia (Gastrointestinal disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastric stenosis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mallory-weiss syndrome (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 25
Neutropenia (Blood and lymphatic system disorders) | 21
Anaemia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Leukopenia (Blood and lymphatic system disorders) | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Infected lymphocele (Infections and infestations) | 4
Infection (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Abdominal wall abscess (Infections and infestations) | 2
Anal abscess (Infections and infestations) | 2
Device related infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Pelvic abscess (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Abdominal infection (Infections and infestations) | 1
Abdominal sepsis (Infections and infestations) | 1
Acute hepatitis C (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cholecystitis inefective (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Colonic abscess (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 1
Parotid abscess (Infections and infestations) | 1
Peritoneal abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Proctitis infectious (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Subdiaphragmatic abscess (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Vulval cellulitis (Infections and infestations) | 1
Hypertension (Vascular disorders) | 16
Embolism venous (Vascular disorders) | 9
Lymphocele (Vascular disorders) | 8
Deep vein thrombosis (Vascular disorders) | 2
Embolism arterial (Vascular disorders) | 2
Lymphoedema (Vascular disorders) | 2
Arterial thrombosis (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Malignant hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Pyrexia (General disorders) | 6
General physical health deterioration (General disorders) | 4
Asthenia (General disorders) | 3
Chest pain (General disorders) | 2
Impaired healing (General disorders) | 2
Death (General disorders) | 1
Fatigue (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 1
Performance status decreased (General disorders) | 1
Headache (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 3
Generalised tonic-clonic seizure (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Acute myocardial infarction (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Calculus ureteric (Renal and urinary disorders) | 1
Glomerulonephritis (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal infarct (Renal and urinary disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Nicotinic acid deficiency (Metabolism and nutrition disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 1
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1
Alanine aminotransferase abnormal (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase abnormal (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase abnormal (Investigations) | 1
General physical condition abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Suicide attempt (Psychiatric disorders) | 2
Bruxism (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Intestinal operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel + Carboplatin (N=1021)
Neutropenia (Blood and lymphatic system disorders) | 485
Anaemia (Blood and lymphatic system disorders) | 333
Thrombocytopenia (Blood and lymphatic system disorders) | 279
Leukopenia (Blood and lymphatic system disorders) | 109
Nausea (Gastrointestinal disorders) | 393
Diarrhoea (Gastrointestinal disorders) | 258
Constipation (Gastrointestinal disorders) | 255
Vomiting (Gastrointestinal disorders) | 230
Abdominal pain (Gastrointestinal disorders) | 221
Stomatitis (Gastrointestinal disorders) | 110
Abdominal pain upper (Gastrointestinal disorders) | 104
Gingival bleeding (Gastrointestinal disorders) | 75
Headache (Nervous system disorders) | 241
Neuropathy peripheral (Nervous system disorders) | 201
Peripheral sensory neuropathy (Nervous system disorders) | 161
Paraesthesia (Nervous system disorders) | 134
Dizziness (Nervous system disorders) | 75
Dysgeusia (Nervous system disorders) | 68
Hypertension (Vascular disorders) | 552
Fatigue (General disorders) | 372
Asthenia (General disorders) | 135
Mucosal inflammation (General disorders) | 110
Pyrexia (General disorders) | 86
Oedema peripheral (General disorders) | 63
Arthralgia (Musculoskeletal and connective tissue disorders) | 261
Myalgia (Musculoskeletal and connective tissue disorders) | 185
Pain in extremity (Musculoskeletal and connective tissue disorders) | 138
Back pain (Musculoskeletal and connective tissue disorders) | 133
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 132
Bone pain (Musculoskeletal and connective tissue disorders) | 52
Alopecia (Skin and subcutaneous tissue disorders) | 442
Rash (Skin and subcutaneous tissue disorders) | 76
Pruritus (Skin and subcutaneous tissue disorders) | 71
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 301
Cough (Respiratory, thoracic and mediastinal disorders) | 94
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 66
Proteinuria (Renal and urinary disorders) | 317
Urinary tract infection (Infections and infestations) | 122
Nasopharyngitis (Infections and infestations) | 83
Upper respiratory tract infection (Infections and infestations) | 60
Platelet count decreased (Investigations) | 93
Weight increased (Investigations) | 77
Decreased appetite (Metabolism and nutrition disorders) | 94
Insomnia (Psychiatric disorders) | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.